CLINICAL TRIAL: NCT01956253
Title: Single Subject Neratinib in Bladder Cancer
Brief Title: Single Subject Neratinib in Bladder Cancer (NRR)
Status: No longer available | Type: Expanded Access
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 13-2526
Record Dates: First submitted 2013-09-25; First posted 2013-10-08 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Bladder Cancer
Keywords: Bladder Cancer; Neratinib; 13-2526
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — neratinib

STUDY DESIGN:
Expanded Access Types: Individual

INTERVENTIONS:
Drug: Neratinib — 240 mg orally once daily

SUMMARY:
This study will be a single subject study to evaluate the efficacy of the HER2 kinase inhibitor, neratinib, in a patient with metastatic bladder cancer harboring a HER2-GRB7 gene fusion.

ELIGIBILITY:
Inclusion Criteria:

* none

Exclusion Criteria:

* none

We have received FDA approval for a single subject Investigational New Drug (IND) Application to treat a specific patient with the HER2 kinase inhibitor neratinib. Therefore there is no inclusion / exclusion criteria.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2013-07; Primary Completion 2013-09 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Kim, MD, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- North Carolina Cancer Hospital (UNC), Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Lineberger Comprehensive Cancer Center — http://cancer.med.unc.edu/